CLINICAL TRIAL: NCT01902173
Title: Phase I/II Study of the Safety and Efficacy of the AKT Inhibitor GSK2141795 in Combination With Dabrafenib and Trametinib in Patients With BRAF Mutant Cancer
Brief Title: Uprosertib, Dabrafenib, and Trametinib in Treating Patients With Stage IIIC-IV Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: GlaxoSmithKline (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-01320; NCI-2013-01320 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SWOG-S1221; S1221 (Other: SWOG); S1221 (Other: CTEP); U10CA180830 (NIH); U10CA180888 (NIH); U10CA032102 (NIH)
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Locally Advanced Malignant Solid Neoplasm; Locally Advanced Melanoma; Metastatic Malignant Solid Neoplasm; Metastatic Melanoma; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7; Unresectable Malignant Solid Neoplasm; Unresectable Melanoma
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasm Metastasis; Melanoma | interventions — Biopsy; Specimen Handling; dabrafenib; Magnetic Resonance Spectroscopy; trametinib; GSK2141795

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (uprosertib, dabrafenib, trametinib) (Experimental): Dabrafenib mesylate and uprosertib (Phase I): Patients receive dabrafenib PO BID and uprosertib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo a CT scan, MRI, and blood sample collection throughout trial. Patients may also undergo a biopsy throughout the trial.
  Dabrafenib mesylate, trametinib dimethyl sulfoxide, and uprosertib (Phase I and Phase II): Patients receive dabrafenib PO BID, trametinib PO QD, and uprosertib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo a CT scan, MRI, and blood sample collection throughout trial. Patients may also undergo a biopsy throughout the trial.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Dabrafenib Mesylate; Procedure: Magnetic Resonance Imaging; Drug: Trametinib Dimethyl Sulfoxide; Drug: Uprosertib

INTERVENTIONS:
Procedure: Biopsy — Undergo a biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo a CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Dabrafenib Mesylate — Given PO
  Other Names: Dabrafenib Methanesulfonate; GSK2118436 Methane Sulfonate Salt; GSK2118436B; Tafinlar
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Trametinib Dimethyl Sulfoxide — Given PO
  Other Names: Mekinist; Meqsel; Spexotras
Drug: Uprosertib — Given PO
  Other Names: GSK2141795; Oral Akt Inhibitor GSK2141795

SUMMARY:
This phase I/II trial studies the side effects and the best dose of uprosertib when given together with dabrafenib and trametinib and to see how well they work in treating patients with stage IIIC-IV cancer. Uprosertib, dabrafenib, and trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving uprosertib with dabrafenib and trametinib may be a better treatment for cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety of dabrafenib mesylate (dabrafenib) in combination with uprosertib (GSK2141795) and select the optimal dose of GSK2141795 for the phase II portion in patients with BRAF mutant cancer. (Effective November 15, 2014, this trial will not proceed to the phase II study of dabrafenib and GSK2141795, but will move to an evaluation of triple therapy). (Phase I) II. To assess the safety of dabrafenib and trametinib dimethyl sulfoxide (trametinib) and GSK2141795 in combination and select the optimal dose of the combination for the phase II portion in patients with BRAF mutant cancer. (Phase I) III. To evaluate the objective response rate (confirmed and unconfirmed, complete and partial responses) in patients with BRAF^V600 mutant metastatic melanoma who have previously progressed on BRAF^V600 inhibitor-based therapy (BRAFi), or BRAFi + MEK inhibitor-based therapy (MEKi). (Phase II)

SECONDARY OBJECTIVES:

I. To estimate overall survival and progression-free survival. II. To assess the toxicity profile of the recommended phase II dose. III. To assess response (complete and partial, confirmed and unconfirmed) of patients enrolled on each phase I portion).

TRANSLATIONAL MEDICINE OBJECTIVES:

I. To explore the molecular mechanisms of acquired resistance to BRAF inhibitor therapy using available biopsies of lesions that progressed during prior BRAF inhibitor-based therapy.

II. To explore potential drug-drug interactions between dabrafenib and GSK2141795 leading to changes in the expected exposure with either agent compared to prior experience. (Phase I)

OUTLINE: This is a phase I, dose-escalation study of uprosertib followed by a phase II study. Dose escalation of dabrafenib mesylate, trametinib dimethyl sulfoxide, and uprosertib will be initiated after completion of the dabrafenib + uprosertib phase I dose escalation.

Dabrafenib mesylate and uprosertib (Phase I): Patients receive dabrafenib orally (PO) twice daily (BID) and uprosertib PO once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo a computed tomography (CT) scan, magnetic resonance imaging (MRI), and blood sample collection throughout trial. Patients may also undergo a biopsy throughout the trial.

Dabrafenib mesylate, trametinib dimethyl sulfoxide, and uprosertib (Phase I and Phase II): Patients receive dabrafenib PO BID, trametinib PO QD, and uprosertib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo a CT scan, magnetic MRI, and blood sample collection throughout trial. Patients may also undergo a biopsy throughout the trial.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* PHASE I PORTION ELIGIBILITY CRITERIA:
* Patients must have BRAF^V600 mutant metastatic cancer irrespective of the histology or prior therapy; BRAF^V600 mutant status must be documented by a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory; use of an Food and Drug Administration (FDA)-approved test is preferred although other BRAF tests at a CLIA-certified laboratory may also be accepted
* Patients must have locally advanced unresectable stage IIIC or metastatic stage IV cancer with either progression to prior therapy or a newly diagnosed cancer that does not have an available treatment with curative intent
* Patients must have a complete physical examination and medical history within 28 days prior to registration
* Patients must have measurable or non-measurable disease; all measurable lesions must be assessed (by physical examination, computed tomography [CT], or magnetic resonance imaging [MRI] scan) within 28 days prior to registration; tests to assess non-measurable disease must be performed within 42 days prior to registration; all disease must be assessed and documented on the baseline tumor assessment form (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1)
* All patients must undergo a CT or MRI of the brain within 42 days prior to registration; patients with asymptomatic brain metastases or previously treated brain metastases that are stable (i.e. not requiring corticosteroids) at the time of registration will be eligible
* Patients may have received prior systemic therapy (chemotherapy, immunotherapy, biologic therapy, or combination regimens); all adverse events associated with prior treatment must have resolved to < grade 1 prior to registration
* Patients progressing on a prior BRAF inhibitor-based therapy will be eligible, as are patients naive to BRAF inhibitor therapy; resistance to BRAF inhibitor-based therapy will be defined as progressive disease by RECIST 1.1 criteria while receiving therapy with a BRAF inhibitor (vemurafenib or dabrafenib, alone or in combination with a mitogen-activated protein kinase [MEK] inhibitor); this may be innate resistance (patients who never achieved a tumor response while on BRAF inhibitor therapy) or acquired resistance (progression after having a tumor response to BRAF inhibitor therapy); there will not be a period of break between progression on the prior BRAF inhibitor-based therapy and the start of dabrafenib, trametinib and GSK2141795
* Patients may have received prior surgery (for both the primary and stage IV disease); all adverse events associated with prior surgery must have resolved to =< grade 1 prior to registration
* Patients may have received prior radiation therapy; all adverse events associated with prior radiation therapy must have resolved to =< grade 1 prior to registration
* Patients must be willing to submit blood for pharmacokinetics; sites must order S1221 pharmacokinetic (PK) kit immediately after registration; the Southwest Oncology Group (SWOG) patient identification (ID) number must be provided on the S1221 PK Kit request form
* Patients must have available and be willing to submit baseline tissue taken at the time of disease progression to prior BRAF inhibitor-based therapy (either fresh frozen [preferred], or paraffin-embedded tumor blocks) OR must have a site of disease that can be biopsied within this study for translational medicine studies; tissue may be from an archival biopsy or a new biopsy after the patient has been registered to the protocol; since patients are referred to this protocol after progression on prior BRAF inhibitor-based therapy, the biopsy taken at the time of progression will be used as the baseline biopsy for this study; patients must be willing to submit plasma and whole blood for translational medicine studies
* Patients must have Zubrod performance status =< 1
* Absolute neutrophil count (ANC) >= 1,200/ul (obtained within 28 days prior to registration)
* Platelets >= 100,000/ul (obtained within 28 days prior to registration)
* Hemoglobin >= 9 g/dL (obtained within 28 days prior to registration)
* Total bilirubin =< 1.5 x institutional upper limit of normal (IULN) (or =< 2.5 x ULN for patients with Gilbert's syndrome) (with 28 days prior to registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x IULN (or < 5 x IULN for patients with known liver metastases) (obtained within 28 days prior to registration)
* Serum albumin >= 2.5 g/dL (obtained within 28 days prior to registration)
* Serum creatinine =< 1.5 mg/dL OR measured or calculated creatinine clearance >= 50 mL/min (obtained within 28 days prior to registration)
* Patient must have a left ventricular ejection fraction >= institutional lower limit of normal (LLN) by echocardiogram (ECHO) or multigated acquisition (MUGA) within 28 days prior to registration
* Patients with melanoma must have a serum lactate dehydrogenase (LDH) test performed within 28 days prior to registration
* Patients with human immunodeficiency virus (HIV) are eligible if they are not on antiviral agents and have adequate cluster of differentiation (CD)4 counts (>= 500 mm^3)
* Patients receiving anticoagulation treatment are allowed to participate with international normalized ratio (INR) established within the therapeutic range
* Women of childbearing potential must have a negative pregnancy test within 14 days of registration
* Patients must be able to retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels; patients who have feeding tubes can enroll in the study provided that the capsules do not need to be modified
* Patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* Patients must be >= 18 years of age
* Patients must have a serum albumin >= 2.5 g/dL within 28 days prior to registration
* PHASE II PORTION ELIGIBILITY CRITERIA:
* Patients must have histologically confirmed melanoma with BRAF^V600 mutation; patients must have stage IIIC or stage IV disease
* Patients must have received prior BRAF inhibitor therapy (e.g. dabrafenib, vemurafenib) within 56 days prior to registration; prior trametinib therapy is permitted; patients are not required to interrupt BRAF or MEK inhibitor therapy prior to the initiation of three agent combination therapy on study
* Patients must have measurable disease; all measurable lesions must be assessed (by physical examination, CT, or MRI scan) within 28 days prior to registration; tests to assess non-measurable disease must be performed within 42 days prior to registration; patients whose only measurable disease is within a previous radiation therapy port must demonstrate clearly progressive disease (in the opinion of the treating investigator) prior to registration; all disease must be assessed and documented on the baseline tumor assessment form (RECIST 1.1)
* Patients must have Zubrod performance status =< 2
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years; patients with history of RAS mutation-positive tumors are not eligible regardless of interval from the current study; Note: Prospective RAS testing is not required; however, if the results of previous RAS testing are known, they must be used in assessing eligibility

Exclusion Criteria:

* Patients must not have a corrected QT (QTc) interval >= 480 msecs within 28 days prior to registration
* Patients must not have a history of acute coronary syndromes (including unstable angina), myocardial infarction within 6 months, coronary angioplasty, or stenting within the past 24 weeks; class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system; or history of known cardiac arrhythmias (such as atrial fibrillation) unless it has been stably controlled for > 30 days prior to registration; abnormal cardiac valve morphology (>= grade 2) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis]) can be entered on study; subjects with moderate valvular thickening are not eligible
* At the time of registration, patients must not be receiving any medications or substances that are strong inhibitors or inducers of cytochrome P450, family 3, subfamily A (CYP3A) or cytochrome P450, family 2, subfamily C, polypeptide 8 (CYP2C8); patients must not be planning to use herbal remedies (e.g., St. John's wort), or strong inhibitors or inducers of P-glycoprotein (Pgp) or breast cancer resistance protein 1 (Bcrp1)
* Patients must not be pregnant or nursing due to unknown teratogenic side effects; women/men of reproductive potential must have agreed to use an effective contraceptive method; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; hormonal contraception is not allowed due to drug interactions which can render hormonal contraceptives ineffective; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Patient must not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, previously diagnosed type 1 diabetes mellitus/type 2 diabetes, psychiatric illness/social situations, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, that would limit compliance with study requirements; patients must not have any evidence of mucosal or internal bleeding; patients must not have a history of pneumonitis or interstitial lung disease; patients must not have received any major surgery within four weeks prior to registration
* Patients must not have an active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Patients must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to dabrafenib or other agents used in this study including dimethyl sulfoxide (DMSO)
* Patients with known history or current evidence of retinal vein occlusion (RVO) are not eligible:

  * History of RVO, or predisposing factors to RVO (e.g. uncontrolled glaucoma or ocular hypertension, uncontrolled systemic disease such as hypertension, diabetes mellitus, or history of hyperviscosity or hypercoagulability syndromes)
  * Visible retinal pathology as assessed by ophthalmic exam that is considered a risk factor for RVO such as:

    * Evidence of new optic disc cupping
    * Evidence of new visual field defects
    * Intraocular pressure > 21 mmHg
    * NOTE: Ophthalmic exam is required for all patients; exam must be obtained within 28 days prior to registration
* Patients must not have uncontrolled hypertension (defined as systolic blood pressure > 140 mm Hg and/or diastolic blood pressure > 90 mm Hg which cannot be controlled by anti-hypertensive therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-10-08 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2023-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Ribas, Principal Investigator — SWOG Cancer Research Network
Locations (16):
- United States (16):
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - PeaceHealth Southwest Medical Center, Vancouver, Washington

REFERENCES:
- [Derived] Algazi AP, Moon J, Lao CD, Chmielowski B, Kendra KL, Lewis KD, Gonzalez R, Kim K, Godwin JE, Curti BD, Latkovic-Taber M, Lomeli SH, Gufford BT, Scumpia PO, Lo RS, Othus M, Ribas A. A phase 1 study of triple-targeted therapy with BRAF, MEK, and AKT inhibitors for patients with BRAF-mutated cancers. Cancer. 2024 May 15;130(10):1784-1796. doi: 10.1002/cncr.35200. Epub 2024 Jan 23. PMID 38261444

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 27 participants were enrolled, however 1 participant on the Dabrafenib + GSK2141795 75 mg arm and 1 participant on the Dabrafenib + Trametinib 1.5mg + GSK2141795 25mg were found to be ineligible. Furthermore, 3 participants on the Dabrafenib + GSK2141795 75 mg arm did not receive protocol treatment were not evaluable for any study endpoint.
Groups:
- Dabrafenib + GSK2141795 50 mg: Doublet regimen cohort 1: participants were given 150 mg of dabrafenib twice daily and 50 mg of GSK2141795 once daily.
- Dabrafenib + GSK2141795 75 mg: Doublet regimen cohort 2: participants were given 150 mg of dabrafenib twice daily and 75 mg of GSK2141795 once daily.
- Dabrafenib + Trametinib 1.5mg + GSK2141795 25mg: Triplet regimen cohort 1: participants were given 150 mg of dabrafenib twice daily, 1.5 mg of trametinib and 25mg of GSK2141795 once daily.
- Dabrafenib + Trametinib 1.5mg + GSK2141795 50mg: Triplet regimen cohort 2: participants were given 150mg of dabrafenib twice daily, 1.5mg of trametinib and 50mg of GSK2141795 once daily.
- Dabrafenib + Trametinib 1.5mg + GSK2141795 75mg: Triplet regimen cohort 3: participants were given 150 mg of dabrafenib twice daily, 1.5 mg of trametinib and 75mg of GSK2141795 once daily.
- Dabrafenib + Trametinib 2.0mg + GSK2141795 75mg: Triplet regimen cohort 4: participants were given 150 mg of dabrafenib twice daily, 2 mg of trametinib and 75 mg of GSK2141795 once daily.
Period: Phase 1 Doublet Regimen Cohort 1
Arm/Group | Dabrafenib + GSK2141795 50 mg | Dabrafenib + GSK2141795 75 mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 25mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 50mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 75mg | Dabrafenib + Trametinib 2.0mg + GSK2141795 75mg
Started | 3 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Progression/relapse | 2 | 0 | 0 | 0 | 0 | 0
Period: Phase 1 Doublet Regimen Cohort 2
Arm/Group | Dabrafenib + GSK2141795 50 mg | Dabrafenib + GSK2141795 75 mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 25mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 50mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 75mg | Dabrafenib + Trametinib 2.0mg + GSK2141795 75mg
Started | 0 | 9 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 9 | 0 | 0 | 0 | 0
Not completed — Progression/relapse | 0 | 5 | 0 | 0 | 0 | 0
Not completed — Ineligible | 0 | 1 | 0 | 0 | 0 | 0
Not completed — No treated | 0 | 3 | 0 | 0 | 0 | 0
Period: Phase 1 Triplet Regimen Cohort 1
Arm/Group | Dabrafenib + GSK2141795 50 mg | Dabrafenib + GSK2141795 75 mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 25mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 50mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 75mg | Dabrafenib + Trametinib 2.0mg + GSK2141795 75mg
Started | 0 | 0 | 4 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 4 | 0 | 0 | 0
Not completed — Progression/relapse | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Ineligible | 0 | 0 | 1 | 0 | 0 | 0
Period: Phase 1 Triplet Regimen Cohort 2
Arm/Group | Dabrafenib + GSK2141795 50 mg | Dabrafenib + GSK2141795 75 mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 25mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 50mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 75mg | Dabrafenib + Trametinib 2.0mg + GSK2141795 75mg
Started | 0 | 0 | 0 | 3 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 3 | 0 | 0
Not completed — Ongoing treatment | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Progression/relapse | 0 | 0 | 0 | 2 | 0 | 0
Period: Phase 1 Triplet Regimen Cohort 3
Arm/Group | Dabrafenib + GSK2141795 50 mg | Dabrafenib + GSK2141795 75 mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 25mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 50mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 75mg | Dabrafenib + Trametinib 2.0mg + GSK2141795 75mg
Started | 0 | 0 | 0 | 0 | 3 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Ongoing | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Progression/relapse | 0 | 0 | 0 | 0 | 2 | 0
Period: Phase 1 Triplet Regimen Cohort 4
Arm/Group | Dabrafenib + GSK2141795 50 mg | Dabrafenib + GSK2141795 75 mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 25mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 50mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 75mg | Dabrafenib + Trametinib 2.0mg + GSK2141795 75mg
Started | 0 | 0 | 0 | 0 | 0 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Progression/relapse | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1
Period: Phase II
Arm/Group | Dabrafenib + GSK2141795 50 mg | Dabrafenib + GSK2141795 75 mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 25mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 50mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 75mg | Dabrafenib + Trametinib 2.0mg + GSK2141795 75mg
Started | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total number of eligible and evaluable patients i.e. patients that received at least one dose of protocol therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabrafenib + GSK2141795 50 mg | Dabrafenib + GSK2141795 75 mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 25mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 50mg | Dabrafenib + Trametinib 1.5mg + GSK2141795 75mg | Dabrafenib + Trametinib 2.0mg + GSK2141795 75mg | Total
Number analyzed (Participants) | 3 | 5 | 3 | 3 | 3 | 5 | 22
Age, Continuous [Median (Full Range); unit: years] | 60.7 [52.0 to 65.8] | 64.4 [40.5 to 70.2] | 63.9 [45.7 to 68.5] | 40.1 [18.5 to 57.5] | 56.7 [28.5 to 70.2] | 50.4 [48.8 to 77.1] | 58.1 [18.5 to 77.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2 | 2 | 2 | 8
  Male | 3 | 4 | 2 | 1 | 1 | 3 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 5 | 3 | 3 | 2 | 5 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 5 | 3 | 3 | 2 | 5 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
Prior BRAF inhibitor [Count of Participants; unit: Participants]
  Yes | 2 | 4 | 1 | 1 | 2 | 3 | 13
  No | 1 | 1 | 2 | 2 | 1 | 1 | 8
  Not reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Type of cancer [Count of Participants; unit: Participants]
  Melanoma | 2 | 4 | 2 | 3 | 3 | 4 | 18
  Lung | 0 | 1 | 1 | 0 | 0 | 1 | 3
  Thyroid | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum-tolerated Dose (MTD) of Akt Inhibitor GSK2141795 in Combination With Dabrafenib.
Description: MTD was evaluated by testing increasing doses up to 75 mg once a day, given in combination with dabrafenib dosed at 150 mg twice daily. MTD reflects the highest dose that did not cause a DLT. DLTs were defined as treatment regimen related: febrile neutropenia; Grade 4 neutropenia lasting more than 7 days; Grade 4 platelet count decrease; Grade 3-4 rash, fever, or hyperglycemia > 14 days, e) Grade 3-4 non-hematologic adverse events lasting greater than 7 days. Adverse events were graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: Every 2 weeks during days 1-56 of treatment.
Population: Eligible, analyzable and evaluable participants that were assessed for DLT. In the Dabrafenib + GSK2141795 75 mg arm, 1 participant was ineligible, 3 participants were not analyzable, and 1 participant did not satisfy protocol-specified criteria for DLT evaluation. These patients were excluded from DLT analysis.
Measure: Number; unit: mg
Groups:
- Phase 1 Doublet Regimen: All analyzable patients who experienced a dose limiting toxicity OR at least received GSK2141795 for 11 days in Cycle 1 and dabrafenib for 28 days in cycles 1 and 2 OR at least received GSK2141795 for 11 days in Cycle 1 and 50% of dabrafenib in Cycle 1
Arm/Group | Phase 1 Doublet Regimen
Number analyzed (Participants) | 7
mg | 75

2. Primary Outcome: Maximum-tolerated Dose (MTD) of Akt Inhibitor GSK2141795 in Combination With Dabrafenib and Trametinib.
Description: MTD was evaluated by testing increasing doses up to 75 mg once a day, given in combination with dabrafenib dosed at 150 mg twice daily and trametinib at either 1.5 mg or 2 mg once a day. MTD reflects the highest dose that did not cause a dose-limiting toxicity (DLT). DLTs were defined as treatment regimen related: febrile neutropenia; Grade 4 neutropenia lasting more than 7 days; Grade 4 platelet count decrease; Grade 3-4 rash, fever, or hyperglycemia > 14 days, e) Grade 3-4 non-hematologic adverse events lasting greater than 7 days. Adverse events were graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
  Note: MTD for the triplet regimen could not be determined due to the end of supply of the study drug. Number reported is the maximum dose of GSK2141795 that was assessed in combination with 150 mg Dabrafenib and 2 mg trametinib.
Time Frame: Every 2 weeks during days 1-56 of treatment.
Population: Eligible and evaluable participants that were assessed for DLT. 1 participant in the Dabrafenib + Trametinib 1.5 mg + GSK2141795 25 mg was not eligible. 1 participant in the Dabrafenib + Trametinib 2.0 mg + GSK2141795 75 mg arm did not satisfy protocol-specified criteria for DLT evaluation and was thus excluded.
Measure: Number; unit: mg
Groups:
- Phase 1 Triplet Regimen: All analyzable patients who experienced a dose limiting toxicity OR at least received GSK2141795 for 11 days in Cycle 1 and dabrafenib and trametinib for 28 days each in cycles 1 and 2 OR at least received GSK2141795 for 11 days in Cycle1 and 50% of dabrafenib and trametinib each in Cycle 1
Arm/Group | Phase 1 Triplet Regimen
Number analyzed (Participants) | 13
mg | 75

3. Primary Outcome: Objective Response Rate (Confirmed and Unconfirmed, Complete and Partial Responses) as Assessed by RECIST Version 1.1 of the Doublet Regimen GSK2141795 + Dabrafenib at the Phase I Determined MTD. (Phase II)
Description: All measurable lesions up to a maximum of 2 lesions per organ 5 lesions in total, representative of all involved organs, were identified as target lesions at baseline. All other lesions (or sites of disease) were identified as non-target lesions.
  Complete Response (CR): Complete disappearance of all target and nontarget lesions. No new lesions. No disease related symptoms. Any lymph nodes (whether target or non-target) must have reduction in short axis to < 1.0 cm.
  Partial Response (PR): <= 30% decrease under baseline of the sum of appropriate diameters of all target measurable lesions. No unequivocal progression of non-measurable disease. No new lesions.
  Unconfirmed CR: One objective status of CR documented before progression or symptomatic deterioration but not qualifying as CR or PR.
  Unconfirmed PR: One objective status of PR documented before progression or symptomatic deterioration but not qualifying as CR, PR or unconfirmed CR.
Time Frame: Disease assessments every 8 weeks for up to 3 years
Population: No participants were enrolled to Phase II portion due to the end of the supply of GSK2141795
Groups:
- Dabrafenib + GSK2141795 at MTD: Patients who received at least one dose of protocol therapy at the Phase I determined MTD.
Arm/Group | Dabrafenib + GSK2141795 at MTD
Number analyzed (Participants) | 0

4. Primary Outcome: Objective Response Rate (Confirmed and Unconfirmed, Complete and Partial Responses) as Assessed by RECIST Version 1.1 of the Triplet Regimen GSK2141795 + Dabrafenib + Trametinib at the Phase I Determined MTD. (Phase II)
Description: as for outcome 3
Time Frame: Disease assessments every 8 weeks for up to 3 years
Population: No participants were enrolled to Phase II portion due to the end of the supply of GSK2141795
Groups:
- Dabrafenib + Trametinib + GSK2141795 at MTD: Patients who received at least one dose of protocol therapy at the Phase I determined MTD.
Arm/Group | Dabrafenib + Trametinib + GSK2141795 at MTD
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival (Phase II) of Patients Treated at the Phase I Determined MTD of Doublet Regimen
Description: Estimated with 95% confidence interval.
Time Frame: From date of registration to date of death due to any cause, assessed up to 3 years
Population: No participants were enrolled to Phase II portion due to the end of the supply of GSK2141795
Groups:
- GSK2141795 + Dabrafenib at the Phase I Determined MTD: Patients who received at least 1 dose of protocol therapy at the Phase I determined MTD
Arm/Group | GSK2141795 + Dabrafenib at the Phase I Determined MTD
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival (Phase II) of Patients Treated at the Phase I Determined MTD of Triplet Regimen
Description: Estimated with 95% confidence interval.
Time Frame: From date of registration to date of death due to any cause, assessed up to 3 years
Population: No participants were enrolled to Phase II portion due to the end of the supply of GSK2141795
Groups:
- GSK2141795 + Dabrafenib + Trametinib at Phase I Determined MTD: Patients who received at least 1 dose of protocol therapy at the Phase I determined MTD
Arm/Group | GSK2141795 + Dabrafenib + Trametinib at Phase I Determined MTD
Number analyzed (Participants) | 0

7. Secondary Outcome: Progression-free Survival as Assessed by RECIST Version 1.1 of the Doublet Regimen at the Phase I Determined MTD (Phase II)
Description: Estimated with 95% confidence interval.
Time Frame: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause, assessed up to 3 years
Population: No participants were enrolled to Phase II portion due to the end of the supply of GSK2141795
Groups:
- Dabrafenib + GSK2141795 at Phase I Determined MTD: Patients who received at least one dose of protocol therapy at the Phase I determined MTD.
Arm/Group | Dabrafenib + GSK2141795 at Phase I Determined MTD
Number analyzed (Participants) | 0

8. Secondary Outcome: Progression-free Survival as Assessed by RECIST Version 1.1 of the Triplet Regimen at the Phase I Determined MTD (Phase II)
Description: Estimated with 95% confidence interval.
Time Frame: as for outcome 7
Population: No participants were enrolled to Phase II portion due to the end of the supply of GSK2141795
Groups:
- Dabrafenib + Trametinib + GSK2141795 at Phase I Determined MTD: Patients who received at least one dose of protocol therapy at the phase I determined MTD
Arm/Group | Dabrafenib + Trametinib + GSK2141795 at Phase I Determined MTD
Number analyzed (Participants) | 0

9. Secondary Outcome: Toxicity Rate of MTD Graded by the NCI CTCAE Version 4.0 (Phase II)
Time Frame: Up to 3 years
Population: No participants were enrolled to the Phase II portion due to the end of the supply of GSK2141795
Groups:
- Dabrafenib + GSK2141795 75 mg: All participants on the Phase II triplet combination of dabrafenib, trametinib and GSK2141795 MTD .
Arm/Group | Dabrafenib + GSK2141795 75 mg
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Pharmacokinetic Parameters
Time Frame: Baseline, pre-dose and 1, 2, 4, and 8 hours on day 15, and pre-dose day 29
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Prevalence of Markers
Description: For binary markers, the prevalence will be able to be estimated and exact binomial confidence interval will be calculated. The association between these categorical markers and clinical outcomes will be explored in a preliminary manner, using Fisher's exact test to compare response and a logrank test to compare Kaplan-Meier estimates of overall survival and progression free survival between marker positive and marker negative groups.
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Dabrafenib + GSK2141795 50 mg: Doublet regimen cohort 1: participants were given 150 mg of dabrafenib twice daily and 50 mg of GK2141795 once daily.
- Dabrafenib + GSK2141795 75 mg: Doublet regimen cohort 2: participants were given 150 mg of dabrafenib twice daily and 75 mg of GK2141795 once daily.
- Dabrafenib + Trametinib 1.5 mg + GSK2141795 25 mg: Triplet regimen cohort 1: participants were given 150 mg of dabrafenib twice daily, 1.5 mg of trametinib and 25 mg of GK2141795 once daily.
- Dabrafenib + Trametinib 1.5 mg + GSK2141795 50 mg: Triplet regimen cohort 2: participants were given 150 mg of dabrafenib twice daily, 1.5 mg of trametinib and 50 mg of GK2141795 once daily.
- Dabrafenib + Trametinib 1.5 mg + GSK2141795 75 mg: Triplet regimen cohort 3: participants were given 150 mg of dabrafenib twice daily, 1.5 mg of trametinib and 75 mg of GK2141795 once daily.
- Dabrafenib + Trametinib 2 mg + GSK2141795 75 mg: Triplet regimen cohort 4: participants were given 150 mg of dabrafenib twice daily, 2 mg of trametinib and 75 mg of GK2141795 once daily.
Arm/Group | Dabrafenib + GSK2141795 50 mg | Dabrafenib + GSK2141795 75 mg | Dabrafenib + Trametinib 1.5 mg + GSK2141795 25 mg | Dabrafenib + Trametinib 1.5 mg + GSK2141795 50 mg | Dabrafenib + Trametinib 1.5 mg + GSK2141795 75 mg | Dabrafenib + Trametinib 2 mg + GSK2141795 75 mg
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/5 | 2/3 | 2/3 | 2/3 | 4/5
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/5 | 2/3 | 1/3 | 1/3 | 5/5
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 3/3 | 3/3 | 3/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabrafenib + GSK2141795 50 mg (N=3) | Dabrafenib + GSK2141795 75 mg (N=5) | Dabrafenib + Trametinib 1.5 mg + GSK2141795 25 mg (N=3) | Dabrafenib + Trametinib 1.5 mg + GSK2141795 50 mg (N=3) | Dabrafenib + Trametinib 1.5 mg + GSK2141795 75 mg (N=3) | Dabrafenib + Trametinib 2 mg + GSK2141795 75 mg (N=5)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fever (General disorders) | 1 | 0 | 0 | 0 | 0 | 3
General disorders and admin site conditions - Other (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Localized edema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 1 | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabrafenib + GSK2141795 50 mg (N=3) | Dabrafenib + GSK2141795 75 mg (N=5) | Dabrafenib + Trametinib 1.5 mg + GSK2141795 25 mg (N=3) | Dabrafenib + Trametinib 1.5 mg + GSK2141795 50 mg (N=3) | Dabrafenib + Trametinib 1.5 mg + GSK2141795 75 mg (N=3) | Dabrafenib + Trametinib 2 mg + GSK2141795 75 mg (N=5)
Anemia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac disorders-Other (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Congenital, familial and genetic disorders - Other (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Eye disorders-Other (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Flashing lights (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 3 | 1 | 1 | 3 | 3
Vomiting (Gastrointestinal disorders) | 2 | 2 | 2 | 2 | 1 | 2
Chills (General disorders) | 1 | 2 | 2 | 0 | 1 | 1
Edema limbs (General disorders) | 2 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 3 | 3 | 3 | 1 | 1 | 3
Fever (General disorders) | 1 | 1 | 2 | 2 | 1 | 2
Flu like symptoms (General disorders) | 1 | 2 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
General disorders and admin site conditions - Other (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Irritability (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 2
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bronchial infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Infections and infestations-Other (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Papulopustular rash (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Injury, poison and procedural complications - Other (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 1 | 1
Creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
INR increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Investigations-Other (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 1 | 1 | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 3
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 2
Weight loss (Investigations) | 2 | 1 | 0 | 0 | 1 | 1
White blood cell decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 3
Anorexia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 2
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 1 | 2
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0 | 1 | 0
Dysphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 2 | 0 | 3
Nervous system disorders-Other (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus pain (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vasovagal reaction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 2
Psychiatric disorders-Other (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal and urinary disorders-Other (Renal and urinary disorders) | 0 | 2 | 1 | 0 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 1 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 1 | 3
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0 | 1 | 1
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vascular disorders-Other (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT01902173/Prot_SAP_000.pdf